CLINICAL TRIAL: NCT01110395
Title: 31P Magnetic Resonance Spectroscopy of Heart
Brief Title: Phosphorous Magnetic Resonance Spectroscopy of Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0533
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR Spectroscopy Post-Heart Transplant (Experimental): Patients post heart transplant getting heart biopsy
  Interventions: Diagnostic Test: MR Spectroscopy

INTERVENTIONS:
Diagnostic Test: MR Spectroscopy — MR spectroscopy of myocardial

SUMMARY:
Heart needs constant supply of energy to continue working. Phosphorus magnetic resonance spectroscopy allows us to measure energy produced in the heart. The purpose of this study is to determine if the energy production is reduced in failing heart.

DETAILED DESCRIPTION:
We will use non-invasive phosphorus magnetic resonance spectroscopy technique to measure creatine kinase (CK) flux in failing heart. The studies will be done on Siemens 3.0T human system. We will recruit subjects with LV dysfunction due to prior anterior wall myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with left ventricular dysfunction

Exclusion Criteria:

* Age < 18, pregnant, history of excessive alcohol use, or any condition (e.g. claustrophobia, a pacemaker) that would prevent him/her from completing the magnetic resonance spectroscopy study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Bashir, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lipskaya TY. Mitochondrial creatine kinase: properties and function. Biochemistry (Mosc). 2001 Oct;66(10):1098-111. doi: 10.1023/a:1012428812780. PMID 11736631
- [Background] Nascimben L, Ingwall JS, Pauletto P, Friedrich J, Gwathmey JK, Saks V, Pessina AC, Allen PD. Creatine kinase system in failing and nonfailing human myocardium. Circulation. 1996 Oct 15;94(8):1894-901. doi: 10.1161/01.cir.94.8.1894. PMID 8873665
- [Background] De Sousa E, Veksler V, Minajeva A, Kaasik A, Mateo P, Mayoux E, Hoerter J, Bigard X, Serrurier B, Ventura-Clapier R. Subcellular creatine kinase alterations. Implications in heart failure. Circ Res. 1999 Jul 9;85(1):68-76. doi: 10.1161/01.res.85.1.68. PMID 10400912
- [Background] Nascimben L, Friedrich J, Liao R, Pauletto P, Pessina AC, Ingwall JS. Enalapril treatment increases cardiac performance and energy reserve via the creatine kinase reaction in myocardium of Syrian myopathic hamsters with advanced heart failure. Circulation. 1995 Mar 15;91(6):1824-33. doi: 10.1161/01.cir.91.6.1824. PMID 7882493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from heart transplant clinic
Groups:
- Transplant: Patients with post-OHT
Period: Overall Study
Arm/Group | Transplant
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Heart Failure: Magnetic Resonance Spectroscopy
Arm/Group | Heart Failure
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: An MR Spectroscopy Showing Signal to Noise Ratio to Determine the Level of Heart Failure
Time Frame: 1-2 days
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MR Spectroscopy Post-Heart Transplant
Number analyzed (Participants) | 15
Ratio | 7 (13.67)
Statistical Analysis 1: Comparison: MR Spectroscopy Post-Heart Transplant; We are unable to provide any further data that has been requested. We have supplied all the data that we can possibly provide because the PI has left the institution and we are unable to contact him. We have no other data; Test type: Other — Bland and Altman; mean + SD — Bland Altman; Bland Altman; Mean + SD = 0.05, Standard Error of Mean 1.96 — We have provided all the information that is available to us. The PI has left the institution and we are unable to contact him. We have no further data to correct the errors; There are no other statistical analysis. We have provided all the information that is available to us. We have no other data available to us because the PI has left the institution and we are unable to contact him
Statistical Analysis 2: Comparison: MR Spectroscopy Post-Heart Transplant; Test type: Other; p < 0.05, Mean + SD

ADVERSE EVENTS:
Time Frame: 1-2 days
Groups:
- Post-Heart Transplant: Patients post heart transplant getting heart biopsy
  MR Spectroscopy: MR spectroscopy for myocardial lipid
Arm/Group | Post-Heart Transplant
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
There were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes